CLINICAL TRIAL: NCT02286128
Title: The Effect of NF-кB Dependent Proinflammation on the Overexpression of Receptor of Advanced Glycation End Products (RAGE) and the Osteogenic Differentiation Defect in the Mesenchymal Stem Cell-isolated From Patients With Type 2 Diabetes
Brief Title: Effect of NF-кB Dependent Proinflammation on Osteogenic Differentiation of the Mesenchymal Stem Cells in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Mattabhorn Phornphutkul, Assistant Professor, Chiang Mai University
Other Study IDs: ChiangMaiU
Record Dates: First submitted 2014-10-28; First posted 2014-11-07 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; RAGE; osteoblast
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and RNA (from peripheral blood-derived mesenchymal stem cells)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-diabetic controls: Age-matched non-diabetic subjects
- Type 2 diabetes: Type 2 diabetes with metformin monotherapy failure

SUMMARY:
This study determines whether NF-кB dependent proinflammatory state found in type 2 diabetes yield to a higher RAGE activation in the mesenchymal stem cell, as well as the effects of the proinflammation on osteoblast differentiation impairment and cellular apoptosis in type 2 diabetic patients. This study will compare non-diabetic control subjects and type 2 diabetic patients with metformin monotherapy failure in the aspect of 1) serum markers for NF-кB dependent proinflammatory state and its intracellular signals, 2) osteogenic differentiation and apoptosis of the mesenchymal stem cells, and 3) serum AGE, RAGE and cellular RAGE activation.

DETAILED DESCRIPTION:
This study aims to explore whether proinflammation in type 2 diabetes is an mechanism underlined higher RAGE activation and osteoblast differentiation defect demonstrated in the MSC of type 2 diabetes, as well as the effects of the proinflammation on cellular differentiation and apoptosis of the MSC. Type 2 diabetes was known to be in proinflammatory state due to NF-кB-dependent cytokine secretion (for example, TNF-α, IL1 and IL6), which in turn contribute to NF-кB upregulation. Because RAGE expression is partly regulated by NF-кB signal, the NF-кB upregulation in proinflammatory state observed in type 2 diabetes may entail RAGE overactivation in this population. Therefore, the proinflammatory state and its correlation to cellular NF-кB-dependent RAGE activation is noteworthy to be determined in the MSC of type 2 diabetes. Furthermore, the effect of proinflammation on differentiation potential and apoptosis of the MSC in type 2 diabetes remains to be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes who has HbA1c higher than 6.5% with metformin monotherapy and age-matched non-diabetes control subjects who signed consent form to be in the study.

Exclusion Criteria:

* Patients who use thiazolidinedione, steroid, immunosuppressive medications, antiresorptive agents or anabolic therapy for osteoporosis.
* Patients with elevated serum creatinine higher than 1.4 in female and 1.5 in male.
* Patients with metastases cancer or hematologic malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 30 non-diabetic control subjects, and 45 type 2 diabetic patients who has HbA1c higher than 6.5% with metformin monotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Correlation between NF-кB dependent-proinflammation markers and osteoblast-specific gene expression in the MSC to measure the effects of NF-кB dependent-proinflammation on differentiation potential toward osteoblast in type 2 diabetes. | 2-4 weeks

SECONDARY OUTCOMES:
Correlation between NF-кB dependent-proinflammation markers and apoptotic marker expression in the MSC to measure effects of NF-кB dependent-proinflammation on cellular apoptosis in type 2 diabetes. | 2-4 weeks
Correlation between NF-кB dependent-proinflammation markers and the expression of RAGE and its downstream signals in the MSC to measure effects of NF-кB dependent-proinflammation on cellular RAGE activation in type 2 diabetes. | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mattabhorn Phornphutkul, M.D, Ph.D, Principal Investigator — Chiang Mai University
Locations (1):
- Mattabhorn Phornputkul, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No